CLINICAL TRIAL: NCT00324948
Title: A Double-Blind, Randomized, 6-Month Evaluation of the Safety and Efficacy of Topical Alprostadil in Hysterectomized Women With Female Sexual Arousal Disorder (FSAD)
Brief Title: Topical Alprostadil for Female Sexual Arousal Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VP Clinical, Vivus, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vivus-FSD-10
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2009-03-10 (Estimated); Status verified 2009-03

CONDITIONS: Sexual Dysfunction, Physiological
Keywords: Female sexual arousal disorder; Female sexual dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Alprostadil

INTERVENTIONS:
Drug: Topical alprostadil (PGE-1)

SUMMARY:
Approximately 300 patients with female sexual arousal disorder who meet eligibility criteria will be enrolled and randomized to receive either active drug or matching placebo. After a two-month, non-treatment period, patients will receive study drug for 6 months and will record information about sexual encounters in a daily diary. Study drug will be applied directly to the genital area 30-60 minutes before initiation of sexual activity. The endpoint of the study is based on the use of a standard measure of sexual function (FSEP).

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, placebo-controlled, parallel-design study involving about 300 women who are 21-60 years of age inclusive, who have undergone a hysterectomy (with or without oophorectomy), and who have a primary diagnosis of FSAD. The diagnosis of FSAD will be made based on a medical and sexual history and confirmed using a structured interview by trained personnel. Study subjects will undergo a 2-month non-treatment run-in period followed by a 6-month period of blinded study therapy. Study drug is applied topically to the genitalia 30-60 minutes prior to initiation of sexual activity. Study subjects will complete several questionnaires at various times during the study and will complete a daily diary. The study endpoint is based on the FSEP and other standard questionnaires, as well as safety and tolerability of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 21-60 who have undergone a hysterectomy
* Have a primary diagnosis of female sexual arousal disorder
* Be willing to comply with all study requirements and visit schedules

Exclusion Criteria:

* Known allergy to alprostadil or product excipients
* Have a genital inflammatory or infectious condition or STD
* Have a significant medical condition that would interfere with the study
* Have received an investigational drug within the prior 30 days

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300
Dates: Start 2004-09; Primary Completion 2006-08 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
FSEP

SECONDARY OUTCOMES:
FSFI
Global assessment
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sam Teichman, MD, Study Director — Vivus Clinical Research Department
Locations (2):
- United States (2):
  - Stanford University School of Medicine-Dept of OB/GYN, Stanford, California
  - Radiant Research, Cincinnati, Ohio